CLINICAL TRIAL: NCT05249140
Title: Finding Treatments for Eating Disorders
Acronym: FED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB21-0472
Record Dates: First submitted 2021-06-21; First posted 2022-02-21 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-06

CONDITIONS: Anorexia in Adolescence
Keywords: Transcranial Magnetic Stimulation; Magnetic Resonance Imaging; Adolescence; Anorexia
MeSH Terms: conditions — Anorexia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Repetitive Transcranial Magnetic Stimulation (Experimental): rTMS parameters are intensity 110% resting motor threshold (RMT), frequency 1Hz, duration = 30 minutes (1800 stimulations), targeting the right DLPFC. To target the dorsolateral prefrontal cortex (DLPFC) for rTMS treatment we will use the traditional method (i.e. the 5cm rule; George et al., 1995, 1996; Herwig et al., 2001, 2003; MacMaster et al., 2019), in which the TMS coil is placed 5 cm anterior to the participant's motor cortex along a line to the nasion. Treatments will occur on weekdays at the same time of day for 4 weeks (20 total).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham Repetitive Transcranial Magnetic Stimulation (Sham Comparator): For the sham rTMS group, a sham coil is used: this sham method does not emit any magnetic field, and therefor does not affect brain activity, but it does produce auditory sensations that is indistinguishable from active rTMS in naïve subjects
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS involves a safe, non-invasive, painless application of a magnetic field over the skull to a target brain area in order to change its activity and function.

SUMMARY:
Currently, Family Based Treatment (FBT) is the leading evidence-based, manualized treatment for adolescents with anorexia nervosa (AN). FBT emphasizes parental involvement in addressing disordered eating by supporting the child in eating and refeeding to achieve a healthy body weight and independent eating. Based on multiple RCTs, 50% of AN patients who receive FBT recover, and those who do not are more likely to develop a chronic illness.

Research demonstrates that weight gain of less than 2.3kg (4.8 pounds) by week 4 of FBT predicts that 75% of adolescents with AN will not achieve weight restoration by the end of treatment. FBT works in part by reducing the avoidance of food and increasing the exposure to food triggers, like the treatment of anxiety disorders and obsessive-compulsive disorder (OCD). Thus, researchers postulate that anxiety may be a negative predictor of FBT treatment outcome in the early phase of FBT. In addition, elevated baseline anxiety has been shown to be associated with poorer outcomes at end of treatment and may also impact the likelihood of early response.

To improve clinical response, we need to develop viable biological treatment targets (i.e., brain areas implicated in anxiety) that could be combined with FBT. Such targets can be defined by 1) initially targeting brain areas that mediate symptoms hindering treatment response (i.e., anxiety), and 2) looking at changes in brain chemistry and function.

Thus, repetitive transcranial magnetic stimulation (rTMS) could be an alternative and promising treatment approach for adolescents with AN who do not respond to Phase 1 of FBT. Using rTMS, we can target the brain areas implicated in anxiety in people with anorexia and modulate that activity to reduce symptoms, and thus, facilitate response to FBT. Several studies have shown the rTMS to the right dorsolateral prefrontal cortex (DLPFC) is effective in reducing anxiety across a range of neuropsychiatric disorders. Therefore, it is possible that stimulating the right DLPFC could facilitate treatment efficacy of FBT in youth with AN. Additional explorations of the connections between, and neurochemistry of, the right DLPFC and those mediating emotion in the brain (e.g., amygdala) could aid in our understanding of the networks impeding effective treatment responses and allow for more tailored, precision targeting with TMS.

DETAILED DESCRIPTION:
norexia nervosa (AN) is a serious psychiatric illness with the highest mortality rate of any other psychiatric disorder. Medical complications from starvation and malnutrition and suicide are the most common cause of death. AN is characterized by a person's fear of gaining weight, becoming fat, and body dissatisfaction, and it has a lifetime prevalence of 0.6 to 2.0% in females. Currently, Family Based Treatment (FBT) is the leading evidence-based, manualized treatment for adolescents with AN. FBT emphasizes parental involvement in addressing disordered eating by supporting the child in eating and refeeding in order to achieve a healthy body weight and independent eating. FBT has been shown to promote rapid weight gain in AN patients in several randomized control trials and reduced hospitalization in AN patients . Based on multiple RCTs, 50% of AN patients who receive FBT recover, and those who do not are more likely to develop a chronic illness.

Research demonstrates that weight gain of less than 2.3kg (4.8 pounds) by week 4 of FBT predicts that 75% of adolescents with AN will not achieve weight restoration by the end of treatment . There continues to be limited empirical research and clinical knowledge about what differentiates those who consistently gain weight and those who do not in the critical window for weight gain in the first month of FBT. FBT works in part by reducing the avoidance of food and increasing the exposure to food triggers, similar to the treatment of anxiety disorders and obsessive-compulsive disorder (OCD). Thus, researchers postulate that anxiety may be a negative predictor of FBT treatment outcome in the early phase of FBT. In addition, elevated baseline anxiety has been shown to be associated with poorer outcomes at end of treatment, and may also impact the likelihood of early response.

While FBT is the first-line treatment for adolescents with AN, response is unfortunately not universal. An understanding of the neurobiology of AN could potentially improve treatment development and response. Unfortunately, the neurobiology of AN is poorly understood, and in turn, neuroscientifically-sound treatments are lacking. In order to improve clinical response, we need to develop viable biological treatment targets (i.e. brain areas implicated in anxiety) that could be combined with FBT. Such targets can be defined by 1) initially targeting brain areas that mediate symptoms hindering treatment response (i.e. anxiety), and 2) looking at changes in brain chemistry and function.

Thus, repetitive transcranial magnetic stimulation (rTMS) could be an alternative and promising treatment approach for adolescents with AN who do not respond to Phase 1 of FBT. rTMS involves a safe, non-invasive, painless application of a magnetic field over the skull to a target brain area in order to change its activity and function. Using rTMS, we can target the brain areas implicated in anxiety in people with anorexia and modulate that activity to reduce symptoms, and thus, facilitate response to FBT. Several studies have shown the rTMS to the right dorsolateral prefrontal cortex (DLPFC) is effective in reducing anxiety across a range of neuropsychiatric disorders. Furthermore, some studies have shown that rTMS is effective in reducing core symptoms of anorexia in adults, however, this has yet to be explored in adolescents. Therefore, it is possible that stimulating the right DLPFC could facilitate treatment efficacy of FBT in youth with AN. Additional explorations of the connections between, and neurochemistry of, the right DLPFC and those mediating emotion in the brain (e.g. amygdala) could aid in our understanding of the networks impeding effective treatment responses and allow for more tailored, precision targeting with TMS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Anorexia Nervosa (AN) by medical and psychiatric assessment at the Calgary Eating Disorder Program.
* English fluency (i.e., able to consent and assent to the study)
* Aged 12 to 18
* Medically stable
* Medications for AN or psychiatric disorders are allowed if the dose has been stable for six weeks with adequate compliance, with a commitment to not change medication/dosage during the trial period. If a medication change occurs, the research team will document this.

Exclusion Criteria:

* Diagnosis of mania or psychosis
* Impediments to TMS or MRI (i.e., braces, having non-MRI compatible metals in the body)
* Diagnosis of Autism Spectrum Disorder
* Diagnosis of post-concussive syndrome
* Plans to move/be unavailable for clinic visits for 6 to 9 months after the start of treatment

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome - Change in anxiety as measured by the Multidimensional Anxiety Scale for Children (MASC-2) from baseline to 6 weeks. | Six weeks
  Change in anxiety as measured by the Multidimensional Anxiety Scale for Children (MASC-2) from baseline to 6 weeks in early non-responders to FBT receiving active rTMS as compared to those receiving sham-rTMS.
Primary Outcome - Number of subjects achieving weight restoration | Six weeks
  Number of early non-responders to FBT who achieve weight restoration (i.e., >95% of expected mean BMI) at the end of active rTMS of the DLPFC treatment as compared to those receiving sham-rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Frank P MacMaster, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
We can share anonymous or aggregated data only upon request.